CLINICAL TRIAL: NCT04367402
Title: COST (COvid STudio) ACTION: Study for the Evaluation of Specific Antibodies Anti Covid-19 Linked to Covid-19 Infection, Symptoms and Genetic Expression of ACE2 Polymorphisms in Patients
Brief Title: COST (COvid STudio) ACTION: Study for the Evaluation of Specific Antibodies Anti Covid-19 Linked to Covid-19 Infection, Symptoms and Genetic Expression of ACE2 Polymorphisms in Patients (COST ACTION)
Acronym: COST ACTION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera San Paolo (Other)
Responsible Party: Principal Investigator, Stefano Centanni, Full Professor, Azienda Ospedaliera San Paolo
Other Study IDs: 2020/ST/057
Record Dates: First submitted 2020-04-17; First posted 2020-04-29 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Symptomatic Patients: Patients who had symptoms related to COVID-19 infection
  Interventions: Other: BioMedomics COVID-19 IgM-IgG Rapid Test
- Health people: Healthy people who never had syntomps related to COVID-19 infection
  Interventions: Other: BioMedomics COVID-19 IgM-IgG Rapid Test
- Asyntomatic Individuals: Asyntomatic people to recruit after the restriction have ended
  Interventions: Other: BioMedomics COVID-19 IgM-IgG Rapid Test

INTERVENTIONS:
Other: BioMedomics COVID-19 IgM-IgG Rapid Test — Qualitative test to aid in the diagnosis of COVID-19 novel coronavirus

SUMMARY:
The aims of this study is to define the genetic bases of COVID-19 related disease heterogeneity in frail population, to carry out a retrospective study on individuals w/wo symptoms to verify the reliability of a prognostic/diagnostic test based on IgM/IgG analysis and on the presence of genetic profiling and to explore the therapeutic potential of the modulation of ACE2 expression.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (> 18 years old)

Exclusion Criteria:

* inability to understand and want;
* mentally incapacitated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sample size: 200 symptomatic patients with no other characteristics; 200 health people with no other characteristics; 200 asymptomatic individuals to recruit after the restrictions have ended with no other characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Retrospective study on individuals with or without symptoms to verify the reliability of a prognostic/diagnostic test based on IgM/IgG analysis. | 6 months
  BioMedomics Rapid IgM-IgG Combined Antibody Test for COVID-19 is immunochromatography based. The test card contains colloidal gold-labeled recombinant novel coronavirus antigen and quality control antibody colloidal gold marker, two detection lines (G and M lines) and one quality control line (C) fixed on a nitrocellulose membrane. When 10 microL of test sample is added to the sample well of the test cassette, the sample will move forward along the test card via capillary action. If the sample contains IgM antibody, the antibody will bind to the colloidal gold-labeled novel coronavirus antigen. The antibody/antigen complex will be captured by the anti-human IgM antibody immobilized on the membrane, forming a red M line and indicating a positive result for the IgM antibody. If the sample contains IgG antibodies, the same thing happens, forming a red G line and indicating a positive result for the IgG antibody. If neither antibody is present, a negative result is displayed.

SECONDARY OUTCOMES:
ACE2 expression in patients with COVID-19 infection | 6 months
  By an in silico analysis, we found 2 missense variants in ACE2 gene annotated at residues 82 (rs766996587) and 355 (rs961360700) involved in PPIs with MAF<0.01. Variants in other residues of the ACE2 may affect protein structure and/or activity/localization, influence the binding of the spike protein and thus the virus ability to enter the respiratory tract.In light of its relevance in cell entry, pharmacological approaches aimed at modulating ACE2 expression, through the modulation of SIRT1 activity in the lung or by selective oligo antisense treatment, should help in counteracting COVID-19 infection. Annotated SNPs evaluation of the TMPRSS2 gene showed 4 exonic common polymorphisms (MAF>1%); of these, rs12329760 is a missense variant in the SRCR domain mediating PPI and ligand binding. Common SNPs are at the 3'UTR, possibly involved in regulating mRNA stability and several rare variants mapped in exons encoding the peptidase domain, potentially affecting protein activity.

CONTACTS AND LOCATIONS:
Locations (1):
- AO San Paolo, Milan, IT, Italy